CLINICAL TRIAL: NCT04071392
Title: Pressure Dynamics in the Non-gravid Uterus: Development of an Intrauterine Pressure Threshold to Confirm Tubal Occlusion After Nonsurgical Permanent Contraception
Brief Title: Development of an Intrauterine Pressure Threshold to Confirm Tubal Occlusion
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Womens Imaging & Intervention (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Principal Investigator, Oregon Health and Science University
Other Study IDs: OHSU IRB 11443
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Sterilization, Female; Fallopian Tube Occlusion
Keywords: hysterosalpingogram (HSG); permanent contraception; tubal occlusion; tubal patency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-Essure Group: Healthy women with history of Essure hysteroscopic permanent contraception.
  Eligible participants will then undergo the HSG imaging study - a standard radiological imaging study to determine that the fallopian tubes are open and free of disease. It also checks the uterine cavity for any abnormalities.
  Interventions: Procedure: Hysterosalpingogram (HSG)
- Control Group: Healthy women with no history of permanent contraception.
  Eligible participants will then undergo the HSG imaging study - a standard radiological imaging study to determine that the fallopian tubes are open and free of disease. It also checks the uterine cavity for any abnormalities.
  Interventions: Procedure: Hysterosalpingogram (HSG)

INTERVENTIONS:
Procedure: Hysterosalpingogram (HSG) — An infusion pump delivered saline via balloon catheter under continuous pressure monitoring. After one minute, investigators withdraw the fluid and recorded volumes in and out. Subjects then undergo hysterosalpingogram (HSG) for evaluation of tubal patency.

SUMMARY:
The overarching goal of this study is to find an alternative method to hysterosalpingogram (HSG) to confirm bilateral tubal occlusion after permanent contraception.

DETAILED DESCRIPTION:
The hystero-(uterus)salpingo-(fallopian tube)graphy (HSG) study is a standard radiological imaging study used to evaluate the internal female reproductive parts, the uterus and fallopian tubes. The tubes are a passage that allows fluid and cells to flow between the body cavity and the uterus. Normally, both tubes are open to this flow, a condition called "tubal patency". If one or both tubes is blocked preventing flow of fluid, this is called "tubal occlusion". If there is tubal patency, as the pressure increases in the uterine cavity, fluid will move through the tubes into the body cavity. If the tubes are occluded, pressure will increase in the uterus but the fluid will not move into the tubes.

The long-term goal is to develop an alternative test to confirm both fallopian tubes are blocked after a non-surgical permanent contraception (sterilization) procedure. Currently tubal patency is determined by HSG.

In this study, the investigators evaluate the potential for alternative diagnostic office tests. The study will evaluate whether uterine pressure measurements can predict tubal patency, or whether the change in volume following intrauterine administration of a fixed volume of saline followed by aspiration predicts tubal patency.

Prior to the instillation of contrast solution, investigators will administer a fixed volume of saline at a constant rate until we reach a volume of 10 ml, or the limit of tolerability for the patient. After a wait of 1 min, they will attempt to aspirate the saline, and measure the difference between fluid in and fluid out. The study will also measure intrauterine pressure during the procedure.

Following the saline test, an HSG is done to assess tubal patency.

This study will evaluate healthy parous women in the late follicular phase and women with a history of Essure permanent contraception.

The investigators hypothesize that women with a history of Essure will have higher uterine pressure, higher volume of fluid recovered, and bilateral tubal occlusion by HSG.

ELIGIBILITY:
Inclusion Criteria:

1. Literate in English
2. Ages 18-50 years
3. No history of infertility, and current regular menstrual cycles occurring every 24-37 days
4. At least one full-term vaginal delivery
5. Not be at risk for pregnancy
6. Be willing to undergo a one month washout period if using the pill, patch or ring, or a three month wash out period if using Depo-Medroxyprogesterone acetate (DMPA)
7. Willing to undergo intrauterine saline infusion followed by a single HSG procedure
8. Able to understand and sign approved study informed consent form
9. Willing to complete a pre-procedure questionnaire

Exclusion Criteria:

1. Currently pregnant as confirmed by positive high-sensitivity urine pregnancy test
2. Currently using an intrauterine device (IUD) or contraceptive implant
3. Hypersensitive to radio-opaque contrast
4. History of cesarean section
5. History of tubal ligation by a method other than Essure® or Adiana
6. History recognized as clinically significant by the investigator, such as symptoms of untreated or recent pelvic infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive age (18-50 years) women in the Portland-metro area with either a history of Essure® hysteroscopic permanent contraception or healthy control participants without history of a permanent contraception procedure.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon consenting and enrollment, subjects will be assigned a unique study identification code that will be used instead of their name, medical record number, or other personally identifying information.
  Data and/or specimens from this study will be kept in a repository and may be shared using the participant's unique study identification code with other investigators for future research.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after publication
Access Criteria: Must have Oregon Health & Science University (OHSU) Institutional Review Board (IRB) approval

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-Essure Group: Healthy women with history of Essure hysteroscopic permanent contraception.
  Eligible participants will then undergo the HSG imaging study - a standard radiological imaging study to determine that the fallopian tubes are open and free of disease. It also checks the uterine cavity for any abnormalities.
  Hysterosalpingogram (HSG): An infusion pump delivered saline via balloon catheter under continuous pressure monitoring. After one minute, investigators withdraw the fluid and recorded volumes in and out. Subjects then undergo hysterosalpingogram (HSG) for evaluation of tubal patency.
- Control Group: Healthy women with no history of permanent contraception.
  Eligible participants will then undergo the HSG imaging study - a standard radiological imaging study to determine that the fallopian tubes are open and free of disease. It also checks the uterine cavity for any abnormalities.
  Hysterosalpingogram (HSG): An infusion pump delivered saline via balloon catheter under continuous pressure monitoring. After one minute, investigators withdraw the fluid and recorded volumes in and out. Subjects then undergo hysterosalpingogram (HSG) for evaluation of tubal patency.
Period: Overall Study
Arm/Group | Post-Essure Group | Control Group
Started | 12 | 12
Completed | 10 | 10
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-Essure Group | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (4.5) | 38.4 (6.1) | 38.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 8 | 8 | 16
  Race/Ethnicity: Hispanic | 1 | 1 | 2
  Race/Ethnicity: Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Intrauterine Fluid Volume Lost
Description: After placement of the hysterosalpingogram catheter, investigators use an infusion pump to deliver normal saline under continuous pressure monitoring until reaching one of the following endpoints: delivery of the entire volume of 10mL (milliliter); a peak pressure of 450mmHg (millimeters of Mercury); or the participant requested the infusion to stop due to intolerable discomfort.
  After one minute, investigators withdraw the delivered fluid through the hysterosalpingogram catheter and record the volume instilled and recovered. They then repeat the procedure using contrast under fluoroscopy to confirm tubal patency or occlusion.
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Post-Essure Group | Control Group
Number analyzed (Participants) | 10 | 10
ml | 2.2 [2.0 to 3.8] | 7.8 [7.4 to 8.4]

2. Secondary Outcome: Tolerance of 10 ml Saline Infusion
Description: After placement of the hysterosalpingogram catheter, investigators use an infusion pump to deliver normal saline under continuous pressure monitoring until reaching one of the following endpoints: delivery of the entire volume of 10mL (milliliter); a peak pressure of 450mmHg (millimeters of Mercury); or the participant requested the infusion to stop due to intolerable discomfort.
  The proportion of participants who tolerated the full 10 ml of infused saline was compared between groups.
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Essure Group | Control Group
Number analyzed (Participants) | 10 | 10
Participants
  Tolerated 10 ml saline | 0 | 5
  Did not tolerate 10 ml saline | 10 | 5

ADVERSE EVENTS:
Time Frame: Per protocol, Adverse Event data were not collected for this study.
Description: Per protocol, Adverse Event data were not collected for this study.
Arm/Group | Post-Essure Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04071392/Prot_SAP_000.pdf